CLINICAL TRIAL: NCT04669054
Title: Hospital Interns Psychological State During the COVID-19 Pandemic
Brief Title: Hospital Interns Psychological State During the COVID-19
Acronym: RESICOV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0665
Record Dates: First submitted 2020-12-14; First posted 2020-12-16 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: COVID 19; Depression; Stress Disorders, Post-Traumatic
Keywords: Hospital interns
MeSH Terms: conditions — COVID-19; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The mental health of the French population in response to covid-19 pandemic is of concern.

Health professionals are prone to more mental disorders due to their direct exposure to the pandemic consequences. Indeed, compared to general population, health care workers face enormous in the current health situation, especially those who may be in contact with suspected or confirmed cases (risk of infection, inadequate protection, loss of control, lack of experience in managing the diseases, overwork, stigma, lack of support). Thus, it seems interesting to describe the psychological state of hospital interns during this pandemic.

ELIGIBILITY:
Inclusion criteria:

* Being a DES intern (Occitanie-Est)
* Being on internship as of November 1, 2020

Exclusion criteria:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Occitanie-Est hospital interns
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Depressive Symptomatology (PHQ-9) | at 5 months (6 months of internship)
  evaluation of the participant depressive symptomatology based on the PHQ-9 scale. The PHQ-9 total score ranges from 0 to 27. A score between 0 and 4 indicates absence of depression; a score between 5 and 9 indicates mild depression; a score between 10 and 14 indicates moderate depression; score between 15 and 19 indicates moderately severe depression and score between 20 and 27 indicates sever depression.
Depressive Symptomatology (PHQ-9) | at inclusion (1 month of internship)
  evaluation of the participant depressive symptomatology based on the PHQ-9 scale. The PHQ-9 total score ranges from 0 to 27. A score between 0 and 4 indicates absence of depression; a score between 5 and 9 indicates mild depression; a score between 10 and 14 indicates moderate depression; score between 15 and 19 indicates moderately severe depression and score between 20 and 27 indicates sever depression.
Depressive Symptomatology (PHQ-9) | at 2 months (3 months of internship)
  evaluation of the participant depressive symptomatology based on the PHQ-9 scale. The PHQ-9 total score ranges from 0 to 27. A score between 0 and 4 indicates absence of depression; a score between 5 and 9 indicates mild depression; a score between 10 and 14 indicates moderate depression; score between 15 and 19 indicates moderately severe depression and score between 20 and 27 indicates sever depression.

SECONDARY OUTCOMES:
Sleep evaluation with the Insomnia Severity Index (ISI) | at inclusion (1 month of internship)
  sleep quality evaluation based on the ISI score. The ISI total score ranges from 0 to 28. A score between 0 and 7 indicates an absence of insomnia; a score between 8 and 14 indicates sub-threshold insomnia; a score between 15 and 21 indicates moderate insomnia and a score between 22 and 28 indicates severe insomnia.
Sleep evaluation with the Insomnia Severity Index (ISI) | at 2 months (3 months of internship)
  sleep quality evaluation based on the ISI score. The ISI total score ranges from 0 to 28. A score between 0 and 7 indicates an absence of insomnia; a score between 8 and 14 indicates sub-threshold insomnia; a score between 15 and 21 indicates moderate insomnia and a score between 22 and 28 indicates severe insomnia.
Sleep evaluation with the Insomnia Severity Index (ISI) | at 5 months (6 months of internship)
  sleep quality evaluation based on the ISI score. The ISI total score ranges from 0 to 28. A score between 0 and 7 indicates an absence of insomnia; a score between 8 and 14 indicates sub-threshold insomnia; a score between 15 and 21 indicates moderate insomnia and a score between 22 and 28 indicates severe insomnia.
Anxiety with the Generalised Anxiety Disorder Assessment (GAD-7) | at inclusion (1 month of internship)
  anxiety evaluation based on the GAD-7 score. The GAD-7 total score ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
Anxiety with the Generalised Anxiety Disorder Assessment (GAD-7) | at 2 months (3 months of internship)
  anxiety evaluation based on the GAD-7 score. The GAD-7 total score ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
Anxiety with the Generalised Anxiety Disorder Assessment (GAD-7) | at 5 months (6 months of internship)
  anxiety evaluation based on the GAD-7 score. The GAD-7 total score ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
Psychological pain assessed with visual analogue scale (VAS) | at inclusion (1 month of internship)
  assessment of the psychological pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Psychological pain assessed with visual analogue scale (VAS) | at 2 months (3 months of internship)
  assessment of the psychological pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Psychological pain assessed with visual analogue scale (VAS) | at 5 months (6 months of internship)
  assessment of the psychological pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Physical pain assessed with visual analogue scale (VAS) | at inclusion (1 month of internship)
  assessment of the physical pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Physical pain assessed with visual analogue scale (VAS) | at 2 months (3 months of internship)
  assessment of the physical pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Physical pain assessed with visual analogue scale (VAS) | at 5 months (6 months of internship)
  assessment of the physical pain. The VAS ranges from 0 (none) to 10 (maximum pain).
Suicidal ideation assessed with visual analogue scale (VAS) | at inclusion (1 month of internship)
  assessment of the suicidal ideation. The VAS ranges from 0 (none) to 10 (maximum ideation).
Suicidal ideation assessed with visual analogue scale (VAS) | at 2 months (3 months of internship)
  assessment of the suicidal ideation. The VAS ranges from 0 (none) to 10 (maximum ideation).
Suicidal ideation assessed with visual analogue scale (VAS) | at 5 months (6 months of internship)
  assessment of the suicidal ideation. The VAS ranges from 0 (none) to 10 (maximum ideation).
Anger assessed with the State Anger Expression Inventory (STAXI - state) | at 2 months (3 months of internship)
  anger assessment with the STAXI state scale. The total score ranges from 0 to 50. The higher the score the higher the anger expression.
Anger assessed with the State Anger Expression Inventory (STAXI - state) | at 5 months (6 months of internship)
  anger assessment with the STAXI state scale. The total score ranges from 0 to 50. The higher the score the higher the anger expression.
Anger assessed with the State Anger Expression Inventory (STAXI - state) | at inclusion (1 month of internship)
  anger assessment with the STAXI state scale. The total score ranges from 0 to 50. The higher the score the higher the anger expression.
Stressful Event Impact (Horowitz scale) | at inclusion (1 month of internship)
  assessement of stressful event impact with the Horowitz scale. The total score ranges from 0 to 45. The higher the score the higher the trauma
Stressful Event Impact (Horowitz scale) | at 2 months (3 months of internship)
  assessement of stressful event impact with the Horowitz scale. The total score ranges from 0 to 45. The higher the score the higher the trauma
Stressful Event Impact (Horowitz scale) | at 5 months (6 months of internship)
  assessement of stressful event impact with the Horowitz scale. The total score ranges from 0 to 45. The higher the score the higher the trauma
Psychotropic drugs use | at inclusion (1 month of internship)
  assessement of the psychotropic drugs use increase
Psychotropic drugs use | at 5 months (6 months of internship)
  assessement of the psychotropic drugs use increase
Psychotropic drugs use | at 2 months (3 months of internship)
  assessement of the psychotropic drugs use increase
Tobacco consumption | at 2 months (3 months of internship)
  assessement of the tobacco consumption increase
Tobacco consumption | at inclusion (1 month of internship)
  assessement of the tobacco consumption increase
Tobacco consumption | at 5 months (6 months of internship)
  assessement of the tobacco consumption increase
Alcohol consumption | at 2 months (3 months of internship)
  assessement of the alcohol consumption increase
Alcohol consumption | at inclusion (1 month of internship)
  assessement of the alcohol consumption increase
Alcohol consumption | at 5 months (6 months of internship)
  assessement of the alcohol consumption increase
Illicit substances use | at inclusion (1 month of internship)
  assessement of the illicit substances use increase
Illicit substances use | at 2 months (3 months of internship)
  assessement of the illicit substances use increase
Illicit substances use | at 5 months (6 months of internship)
  assessement of the illicit substances use increase

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC